CLINICAL TRIAL: NCT01506193
Title: Immunogenicity and Safety Study of GlaxoSmithKline Biological's Live Attenuated Measles Mumps Rubella Varicella Vaccine (PriorixTetra™) When Co-administered With Conjugated Meningococcal C Vaccine (Meningitec®, Nuron Biotechs' Vaccine) in Healthy Children
Brief Title: Immunogenicity and Safety Study of PriorixTetra™ When Co-administered With Conjugated MenC Vaccine in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 115555; 2011-001608-37 (EudraCT Number)
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2017-06

CONDITIONS: Rubella; Varicella; Measles; Mumps
Keywords: safety; healthy; conjugated; immunogenicity; children; MenC vaccine; MMRV vaccine
MeSH Terms: conditions — Rubella; Chickenpox; Measles; Mumps | interventions — measles, mumps, rubella, varicella vaccine; MenC-CRM vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Subjects in this arm will receive MMRV vaccine at Visit 1 (Day 0) and MenC vaccine at Visit 2 (Days 35-49).
  Interventions: Biological: PriorixTetra™; Biological: Meningitec
- Group B (Experimental): Subjects will receive MMRV vaccine and MenC vaccine at Visit 1 (Day 0).
  Interventions: Biological: PriorixTetra™; Biological: Meningitec
- Group C (Active Comparator): Subjects will receive Men C vaccine at Visit 1 (Day 0) and MMRV vaccine at Visit 2 (Day 35-49).
  Interventions: Biological: PriorixTetra™; Biological: Meningitec

INTERVENTIONS:
Biological: PriorixTetra™ — One dose administered subcutaneously
  Other Names: MMRV vaccine (GSK208136)
Biological: Meningitec — One dose administered intramuscularly
  Other Names: MenC vaccine

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of GSK Biologicals' investigational measles, mumps, rubella and varicella (MMRV) vaccine (GSK208136, PriorixTetra™) when co-administered along with conjugated Meningococcal C (MenC) vaccine (Meningitec®, Nuron Biotechs' Vaccine) in healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representatives (LAR) can and will comply with the requirements of the protocol.
* A male or female between, and including, 13 and 15 months of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/ LAR of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol starting 30 days prior to the study vaccination/s and ending 42 days after the vaccination/s (at Visit 2), with the exception of inactivated influenza (flu) vaccine, which may be given at any time during the study, including the day of study vaccination/s.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous vaccination against measles, mumps, rubella, varicella/ herpes zoster and/or N. meningitidis serogroup C.
* History of measles, mumps, rubella, varicella and/or N. meningitidis serogroup C diseases.
* Known exposure to measles, mumps, rubella and or varicella starting 30 days prior to enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* Acute disease and/or fever at the time of enrollment.
* Documented human immunodeficiency virus (HIV) positive subject.
* Any contraindications as stated in the Summary of Product Characteristics.
* Administration of immunoglobulins and/or any blood products within three months prior to the first vaccine dose or planned administration during the study period.

Ages: 13 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 716 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2014-02-17 (Actual); Study Completion 2014-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Italy (12):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Chiavari, Liguria
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Cuneo, Piedmont
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Alghero (SS), Sardinia
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Modica (RG), Sicily
  - GSK Investigational Site, Ragusa (RG), Sicily

REFERENCES:
- [Derived] Durando P, Esposito S, Bona G, Cuccia M, Desole MG, Ferrera G, Gabutti G, Pellegrino A, Salvini F, Henry O, Povey M, Marchetti F. The immunogenicity and safety of a tetravalent measles-mumps-rubella-varicella vaccine when co-administered with conjugated meningococcal C vaccine to healthy children: A phase IIIb, randomized, multi-center study in Italy. Vaccine. 2016 Aug 5;34(36):4278-84. doi: 10.1016/j.vaccine.2016.07.009. Epub 2016 Jul 14. PMID 27423382

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Priorix-Tetra + Meningitec Group: Healthy male or female subjects between 13 to 15 months of age who received Meningitec® vaccine co-administered along with Priorix-Tetra™ vaccine at Visit 1 (Day 0). Priorix-Tetra™ vaccine was administered subcutaneously in the deltoid region of the left arm and Meningitec® vaccine was administered intramuscularly in the tricep of the right arm.
- Priorix-Tetra Group: Healthy male or female subjects between 13 to 15 months of age who received Priorix-Tetra™ vaccine at Visit 1 (Day 0) and Meningitec® vaccine at Visit 2 (Days 35-49). Priorix-Tetra™ vaccine was administered subcutaneously in the deltoid region of the left arm and Meningitec® vaccine was administered intramuscularly in the tricep of the right arm.
- Meningitec Group: Healthy male or female subjects between 13 to 15 months of age who received Meningitec® vaccine at Visit 1 (Day 0) and Priorix-Tetra™ vaccine at Visit 2 (Days 35-49). Priorix-Tetra™ vaccine was administered subcutaneously in the deltoid region of the left arm and Meningitec® vaccine was administered intramuscularly in the tricep of the right arm.
Period: Overall Study
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group | Meningitec Group
Started | 351 | 183 | 182
Completed | 337 | 179 | 168
Not Completed | 14 | 4 | 14
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Migrated/moved from study area | 0 | 0 | 1
Not completed — Adverse event, non-fatal | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 8
Not completed — Lost to Follow-up | 8 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group | Meningitec Group | Total
Number analyzed (Participants) | 351 | 183 | 182 | 716
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.4 (0.6) | 13.4 (0.6) | 13.4 (0.7) | 13.4 (0.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 85 | 88 | 340
  Male | 184 | 98 | 94 | 376

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Measles, Mumps, Rubella, and Varicella Virus
Description: Seroconversion was defined as the appearance of antibodies (i.e. concentration/titer ≥ the cut-off value) in the serum of subjects seronegative before vaccination. The cut-off values for serocoversion were 150 mIU/mL, 231 U/mL, 4 IU/mL and 25 mIU/mL for measles, mumps, rubella and varicella, respectively.
Time Frame: At 42 days after vaccination
Population: The analysis was performed on all eligible subjects with post-dose 1 serology results available for at least one antigen in this analysis, included in the ATP cohort for immunogenicity post-dose 1, who received medication/vaccine and who had no underlying medical condition forbidden in the protocol before the Visit 2 last blood draw.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group
Number analyzed (Participants) | 309 | 164
Participants
  Anti-measles ≥ 150 mIU/mL: number analyzed (Participants) | 307 | 163
  Anti-measles ≥ 150 mIU/mL | 305 | 162
  Anti-mumps ≥ 231 U/ML: number analyzed (Participants) | 309 | 162
  Anti-mumps ≥ 231 U/ML | 292 | 151
  Anti-rubella ≥ 4 IU/mL | 309 | 164
  Anti-varicella ≥ 25 mIU/mL: number analyzed (Participants) | 300 | 159
  Anti-varicella ≥ 25 mIU/mL | 299 | 159
Statistical Analysis 1: Comparison: Priorix-Tetra + Meningitec Group vs Priorix-Tetra Group; Immune response for anti-measles antibodies Non-inferiority of Priorix-Tetra™ vaccine co-administered with Meningitec® conjugate vaccine compared to the first dose of Priorix-Tetra™ vaccine alone with respect to anti-measles seroconversion rates (SCRs) at Day 42 after dose 1; Test type: Non-Inferiority or Equivalence — Non-inferiority with respect to seroconversion rates for measles was concluded if the lower limit of the 95% CI around the difference in seroconversion rates between groups would be [-10%] or higher; Difference in percentage = -0.04, 95% CI 2-sided [-1.82 to 2.78]
Statistical Analysis 2: Comparison: Priorix-Tetra + Meningitec Group vs Priorix-Tetra Group; Immune response for anti-mumps antibodies Non-inferiority of Priorix-Tetra™ vaccine co-administered with Meningitec® conjugate vaccine compared to the first dose of Priorix-Tetra™ vaccine alone with respect to anti-mumps seroconversion rates (SCRs) at Day 42 after dose 1; Test type: Non-Inferiority or Equivalence — Non-inferiority with respect to seroconversion rates for mumps was concluded if the lower limit of the 95% CI around the difference in seroconversion rates between groups would be [-10%] or higher; Difference in percentage = 1.29, 95% CI 2-sided [-3.04 to 6.67]
Statistical Analysis 3: Comparison: Priorix-Tetra + Meningitec Group vs Priorix-Tetra Group; Immune response for anti-rubella antibodies Non-inferiority of Priorix-Tetra™ vaccine co-administered with Meningitec® conjugate vaccine compared to the first dose of Priorix-Tetra™ vaccine alone with respect to anti-rubella seroconversion rates (SCRs) at Day 42 after dose 1; Test type: Non-Inferiority or Equivalence — Non-inferiority with respect to seroconversion rates for rubella was concluded if the lower limit of the 95% CI around the difference in seroconversion rates between groups would be [-10%] or higher; Difference in percentage = 0, 95% CI 2-sided [-1.23 to 2.29]
Statistical Analysis 4: Comparison: Priorix-Tetra + Meningitec Group vs Priorix-Tetra Group; Immune response for anti-varicella antibodies Non-inferiority of Priorix-Tetra™ vaccine co-administered with Meningitec® conjugate vaccine compared to the first dose of Priorix-Tetra™ vaccine alone with respect to anti-varicella seroconversion rates (SCRs) at Day 42 after dose 1; Test type: Non-Inferiority or Equivalence — Non-inferiority with respect to seroconversion rates for varicella was concluded if the lower limit of the 95% CI around the difference in seroconversion rates between groups would be [-10%] or higher; Difference in percentage = -0.33, 95% CI 2-sided [-1.87 to 2.03]

2. Primary Outcome: Number of Seroprotected Subjects for rSBA-MenC Antibodies
Description: Seroprotection was defined as the appearance of rSBA-MenC antibody titer ≥ 1:8.
Time Frame: At 42 days after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra + Meningitec Group | Meningitec Group
Number analyzed (Participants) | 291 | 143
Participants | 286 | 142
Statistical Analysis 1: Comparison: Priorix-Tetra + Meningitec Group vs Meningitec Group; Immune response for rSBA-MenC antibodies Non-inferiority of Meningitec® conjugate vaccine co-administered with Priorix-Tetra™ compared to Meningitec® conjugate vaccine alone with respect to rabbit complement serum bactericidal assay (rSBA-MenC) antibody seroprotection rates (SPRs) at Day 42 after vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority with respect to seroresponse for rSBA-MenC was concluded if the lower limit of the 95% CI around the difference in seroprotection rates between groups would be [-10%] or higher; Difference in percentage = -1.02, 95% CI 2-sided [-3.39 to 2.24]

3. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = Cried when limb is moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site. This outcome measure concerns subjects in Priorix-Tetra + Meningitec Group and Priorix-Tetra Group only. Subjects in Priorix-Tetra Group did not receive Meningitec® vaccine.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with study vaccine administered, on subjects with their symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group
Number analyzed (Participants) | 337 | 177
Participants
  Any Pain, Meningitec: number analyzed (Participants) | 336 | 0
  Any Pain, Meningitec | 79 |
  Grade 3 Pain, Meningitec: number analyzed (Participants) | 336 | 0
  Grade 3 Pain, Meningitec | 4 |
  Any Pain, Priorix-Tetra | 78 | 31
  Grade 3 Pain, Priorix-Tetra | 1 | 1
  Any Redness, Meningitec: number analyzed (Participants) | 336 | 0
  Any Redness, Meningitec | 100 |
  Grade 3 Redness, Meningitec: number analyzed (Participants) | 336 | 0
  Grade 3 Redness, Meningitec | 9 |
  Any Redness, Priorix-Tetra | 92 | 41
  Grade 3 Redness, Priorix-Tetra | 4 | 1
  Any Swelling, Meningitec: number analyzed (Participants) | 336 | 0
  Any Swelling, Meningitec | 68 |
  Grade 3 Swelling, Meningitec: number analyzed (Participants) | 336 | 0
  Grade 3 Swelling, Meningitec | 9 |
  Any Swelling, Priorix-Tetra | 47 | 20
  Grade 3 Swelling, Priorix-Tetra | 1 | 2

4. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability/fussiness and loss of appetite. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal activity. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 15-day (Days 0-14) post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 336 | 177 | 171
Participants
  Any Drowsiness | 148 | 89 | 56
  Grade 3 Drowsiness | 16 | 12 | 6
  Related Drowsiness | 128 | 67 | 46
  Any Irritability/Fussiness | 187 | 104 | 84
  Grade 3 Irritability/Fussiness | 30 | 13 | 7
  Related Irritability/Fussiness | 158 | 82 | 64
  Any Loss of appetite | 178 | 99 | 60
  Grade 3 Loss of appetite | 25 | 12 | 5
  Related Loss of appetite | 138 | 75 | 43

5. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were Parotid / salivary gland swelling and suspected signs of meningism / febrile convulsions. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 parotid / salivary gland swelling = swelling with accompanying general symptoms and Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 336 | 177 | 171
Participants
  Any Parotid / salivary gland swelling | 3 | 4 | 0
  Grade 3 Parotid / salivary gland swelling | 0 | 0 | 0
  Related Parotid / salivary gland swelling | 3 | 3 | 0
  Any Suspected signs of meningism | 1 | 0 | 1
  Grade 3 Suspected signs of meningism | 0 | 0 | 0
  Related Suspected signs of meningism | 1 | 0 | 0

6. Secondary Outcome: Number of Subjects Reporting Fever Per Half Degree
Description: Any fever = fever ≥ 38.0°C on rectal setting, grade 3 fever = fever > 39.5 °C and related = fever assessed by the investigator as causally related to study vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 336 | 177 | 171
Participants
  Any temperature | 159 | 86 | 46
  Grade 3 temperature | 15 | 9 | 4
  Related temperature | 178 | 84 | 28

7. Secondary Outcome: Number of Subjects Reporting Any, Localised and Generalised Rashes
Description: Rash/exanthem was defined as: 1) measles/ rubella rashes (macular or maculo-papular rashes): presence of macules, discolored small patches or spots of the skin, neither elevated nor depressed below the skin's surface. 2) varicella rash (maculo-papulo-vesicular): simultaneous presence of macules, papules and vesicles raised above the skin's surface or other types of rash (heat rash, diaper rash etc.). Any rash = no lesions and grade 3 = > 150 lesions.
Time Frame: Within the 43-day (Days 0-42) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with study vaccine administered, on subjects with their symptom sheets for rash completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 337 | 177 | 171
Participants
  Any, Localised or generalised rash | 91 | 41 | 15
  Any, With fever rash | 59 | 30 | 2
  Any, Varicella like rash | 6 | 1 | 1
  Any, Measles/Rubella like rash | 40 | 16 | 2
  Any, Grade 3 rash | 2 | 1 | 2
  Any, Related rash | 66 | 22 | 6
  Localised, Any rash | 43 | 13 | 9
  Localised, Administration site rash | 3 | 1 | 3
  Localised, Other site rash | 40 | 12 | 6
  Localised, With fever rash | 23 | 10 | 1
  Localised, Varicella like rash | 2 | 0 | 0
  Localised, Measles/Rubella like rash | 15 | 3 | 2
  Localised, Grade 3 rash | 0 | 0 | 1
  Localised, Related rash | 31 | 4 | 6
  Generalised, Any rash | 54 | 28 | 6
  Generalised, With fever rash | 38 | 20 | 1
  Generalised, Varicella like rash | 4 | 1 | 1
  Generalised, Measles/Rubella like rash | 25 | 13 | 0
  Generalised, Grade 3 rash | 2 | 1 | 1
  Generalised, Related rash | 39 | 18 | 0

8. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product reported in addition to those solicited during the clinical study. Any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 43 days (Days 0-42) after each vaccination
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 351 | 183 | 182
Participants | 97 | 61 | 41

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout study period (from Day 0 to approximately Month 4)
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group | Meningitec Group
Number analyzed (Participants) | 351 | 183 | 182
Participants | 6 | 4 | 2

10. Secondary Outcome: Antibody Titers Against Measles, Mumps, Rubella and Varicella Viruses
Description: Antibody titers were summarized by geometric mean concentrations (GMCs) with their 95% confidence intervals (CIs) for the following cut-offs: ≥ 150 mIU/mL, ≥ 231 U/mL, ≥ 4 IU/mL and ≥ 25 mIU/mL for anti-measles, anti-mumps, anti-rubella and anti-varicella, respectively.
Time Frame: At Day 42 after vaccination
Population: The analysis was performed on the ATP cohort for immunogenicity post-dose 1 which included all eligible subjects with post-dose 1 serology results available for at least one antigen, who received medication/vaccine and who had no underlying medical condition forbidden in the protocol before the Visit 2 last blood drawn.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group
Number analyzed (Participants) | 309 | 164
Titers
  Anti-measles: number analyzed (Participants) | 307 | 163
  Anti-measles | 2943.6 [2691.5 to 3219.2] | 3158.5 [2749.7 to 3628]
  Anti-mumps: number analyzed (Participants) | 309 | 162
  Anti-mumps | 1530.7 [1368.4 to 1712.1] | 1591.3 [1346.2 to 1881]
  Anti-rubella | 40.2 [37.3 to 43.3] | 44.9 [40.6 to 49.6]
  Anti-varicella: number analyzed (Participants) | 300 | 159
  Anti-varicella | 156.3 [143.9 to 169.8] | 145.2 [129.5 to 162.8]

ADVERSE EVENTS:
Time Frame: Solicited local & general symptoms: during Days 0-3 and Days 0-14 post-vaccination period, respectively; Unsolicited AEs: during the 43 day (Days 0-42) post each vaccination; SAEs: throughout the entire study period (from Day 0 to approximately Month 4).
Description: The number of occurrences reported for serious adverse events were not available for posting. The number of subjects affected by each specific event was indicated as the number of occurrences.
Arm/Group | Priorix-Tetra + Meningitec Group | Priorix-Tetra Group | Meningitec Group
Serious Adverse Events (participants affected / at risk) | 6/351 | 4/183 | 2/182
Other Adverse Events (participants affected / at risk) | 327/351 | 158/183 | 146/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Priorix-Tetra + Meningitec Group (N=351) | Priorix-Tetra Group (N=183) | Meningitec Group (N=182)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Priorix-Tetra + Meningitec Group (N=351) | Priorix-Tetra Group (N=183) | Meningitec Group (N=182)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 10 (10) | 5 (5)
Somnolence (Nervous system disorders) | 148 (148) | 89 (89) | 56 (56)
Injection site pain (General disorders) | 92 (92) | 31 (31) | 0 (0)
Injection site swelling (General disorders) | 79 (79) | 20 (20) | 1 (1)
Injection site erythema (General disorders) | 121 (121) | 41 (41) | 0 (0)
Decreased appetite (General disorders) | 178 (178) | 99 (99) | 60 (60)
Irritability postvaccinal (General disorders) | 187 (187) | 104 (104) | 84 (84)
Pyrexia (General disorders) | 220 (220) | 114 (114) | 64 (64)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 10 (10) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 91 (91) | 41 (41) | 15 (15)
Pharyngitis (Infections and infestations) | 16 (16) | 10 (10) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.